CLINICAL TRIAL: NCT04230941
Title: Mitigating Cancer-Related Cognitive Impairment in Older Adults With Breast Cancer Receiving Chemotherapy: Memory and Attention Adaptation Training-Geriatrics (MAAT-G) Phase I
Brief Title: Memory and Attention Adaptation Training-Geriatrics (MAAT-G)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Allison Magnuson, Associate Professor of Medicine, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCS19102; 1K76AG064394-01 (NIH)
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Results first posted 2023-07-19 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Cancer-related Problem/Condition; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Usability
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAAT-G Intervention (Experimental): MAAT-G Workshops & participant workbook use (8 workshops)
  Interventions: Behavioral: MAAT-G

INTERVENTIONS:
Behavioral: MAAT-G — Memory and Attention Adaptation Training (MAAT) is a cognitive-behavioral therapy (CBT)-based intervention for CRCD. As a CBT-based intervention, MAAT focuses on an individual's psychological response to injury as compared to the biological events triggering CRCD. MAAT is a series of manualized workshops delivered by a psychologist via video-conferencing, supplemented by a participant workbook, which provide instruction and practice with adaptive behavioral coping skills, stress management techniques, and compensation strategies. MAAT-G has been adapted to optimize usability. We are now testing the feasibility of MAAT-G in older cancer survivors with Mild Cognitive Impairment.

SUMMARY:
Cancer-related cognitive dysfunction (CRCD) affects up to 75% of patients receiving chemotherapy and older adults are at greater risk of developing CRCD, which can negatively affect their functional independence and quality of life. Memory and Attention Adaptation Training (MAAT) is a promising treatment for CRCD that improves perceived cognition in younger cancer survivors, but needs to be adapted for older adults to address their unique needs. The proposed study will adapt MAAT for older adults using feedback from key stakeholders (older adults with cancer and their caregivers), and test usability of the intervention.

DETAILED DESCRIPTION:
Cancer-related cognitive dysfunction (CRCD) is a significant problem, affecting up to 75% of patients receiving chemotherapy. Older adults are at greater risk of developing CRCD which can negatively affect their functional independence and quality of life. Memory and Attention Adaptation Training (MAAT) is a promising tool that improves perceived cognition in younger cancer survivors with CRCD. For older adults with cancer, MAAT could be delivered alongside chemotherapy to mitigate the development of CRCD (when risk is highest) and CRCD-related effects on functional independence for older adults. However, MAAT will require adaptation to meet the unique needs of older adults to optimize usability and efficacy for this population. The overarching goal of this project is to adapt MAAT for older adults using input from patient and caregiver stakeholders (phase I), and subsequently gather data on the preliminary effects of the adapted MAAT (MAAT-Geriatrics [G]) on perceived cognition, objective cognitive measures and functional independence. The provided details pertain to Phase I of the study, which will focus on the adaptation process and usability testing.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Have a diagnosis of invasive breast cancer
2. Planned to receive systemic therapy for breast cancer or actively receiving systemic therapy for breast cancer with two additional cycles remaining.
3. Be age 65 or older
4. Able to provide informed consent
5. Able to read and understand English (or possess a designated health care proxy that can do the same that was designated prior to the patient losing decision-making capabilities)

Patient Exclusion Criteria:

1. Have surgery planned within 3 months of consent
2. Patients who do not have decision-making capacity (decisionally or cognitively impaired) AND do NOT have a previously designated health care proxy (established prior to their cognitive impairment) available to sign consent
3. Patients with breast cancer receiving endocrine therapy as their only systemic therapy will not be eligible.

Eligible Caregiver Inclusion Criteria:

1. Selected by the patient when asked if there is a "family member, partner, friend or caregiver [age 21 or older] with whom you discuss or who can be helpful in health-related matters;" patients who cannot identify such a person ("caregiver") will remain eligible for the study.

Eligible Caregiver Exclusion Criteria:

1. Caregivers unable to understand the consent form due to cognitive, health or sensory impairment will be excluded

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Magnuson, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- MAAT-G Intervention: MAAT-G Workshops & participant workbook use (10 workshops)
  MAAT-G: Memory and Attention Adaptation Training-Geriatrics (MAAT-G) is a cognitive-behavioral therapy (CBT)-based intervention for Cancer Related Cognitive Decline (CRCD). As a CBT-based intervention, MAAT-G focuses on an individual's psychological response to injury as compared to the biological events triggering CRCD. MAAT-G is a series of manualized workshops delivered by a psychologist via video-conferencing, supplemented by a participant workbook, which provide instruction and practice with adaptive behavioral coping skills, stress management techniques, and compensation strategies. MAAT-G has been adapted to optimize usability. We are evaluating the usability of MAAT-G.
- Caregiver: Optional for caregiver to enroll with patient. Caregivers were not required to enroll for patients to be able to participate.
Period: Overall Study
Arm/Group | MAAT-G Intervention | Caregiver
Started | 4 | 1
Completed | 4 (Enrollment paused for usability testing (2021). Usability testing met pre-established threshold (2021). Usability testing now determined complete (2022).) | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MAAT-G Intervention: MAAT-G Workshops & participant workbook use (10 workshops)
  MAAT-G: Memory and Attention Adaptation Training-Geriatrics (MAAT-G) is a cognitive-behavioral therapy (CBT)-based intervention for CRCD. As a CBT-based intervention, MAAT-G focuses on an individual's psychological response to injury as compared to the biological events triggering CRCD. MAAT-G is a series of manualized workshops delivered by a psychologist via video-conferencing, supplemented by a participant workbook, which provide instruction and practice with adaptive behavioral coping skills, stress management techniques, and compensation strategies. MAAT-G has been adapted to optimize usability. We are evaluating the usability of MAAT-G.
- Caregiver: Caregivers were optional to enroll with patients. A caregiver was not required to enroll for a patient to participate.
- Total: Total of all reporting groups
Arm/Group | MAAT-G Intervention | Caregiver | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Full Range); unit: years] | 73.25 [67 to 77] | 78 [78 to 78] | 73.8 [67 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: System Usability Scale (SUS)
Description: The System Usability Scale is a metric to evaluate the usability of the intervention (Patients) and is scored 0 (minimum) to 100 (maximum). Higher scores indicate greater usability. A mean score >68 is consisted with optimal usability.
Time Frame: Post-Intervention (up to 2 weeks)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | MAAT-G Intervention
Number analyzed (Participants) | 4
score on a scale | 90.6 [67.5 to 100]

2. Primary Outcome: Experience Interview
Description: Semi-structured interview with patients and caregivers about experience with MAAT-G. (Patients and caregivers) Qualitative Analysis of transcripts from participant/caregiver interviews will be analyzed for themes on intervention benefit and barriers and facilitators.
Time Frame: Post-Intervention (up to 2 weeks)
Population: MAX QDA Software utilized for qualitative analysis coding
Measure: Count of Participants; unit: Participants
Arm/Group | MAAT-G Intervention | Caregiver
Number analyzed (Participants) | 4 | 1
Participants
  Number of participants describing the MAAT-G intervention as beneficial | 4 | 1
  Number of participants using study-based facilitators to overcome Telehealth barriers | 3 | 1

ADVERSE EVENTS:
Time Frame: From initiation of the intervention to post-assessment time point (approximately 14 weeks).
Groups:
- Caregiver: Caregiver was allowed to enroll with patient. Caregiver enrollment was not required for patient to participate
Arm/Group | MAAT-G Intervention | Caregiver
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 0/4 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT04230941/Prot_SAP_000.pdf